CLINICAL TRIAL: NCT06577883
Title: Chest X-ray Tomosynthesis for Detection of Lung Cancer and Lung Disease
Brief Title: Next Generation Chest X-Ray Tomosynthesis for Screening of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: AIxSCAN, Inc. (Unknown)
Responsible Party: Principal Investigator, Albert Hsiao, Professor in Residence, Department of Radiology, University of California, San Diego
Other Study IDs: 805210
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest X-ray Tomosynthesis Participants: Participants who had a recent, routine clinical chest computed tomography scan for lung cancer screening or evaluation of nodule suspicious for lung cancer will undergo an additional chest X-ray tomosynthesis scan.
  Interventions: Diagnostic Test: Chest X-ray Tomosynthesis

INTERVENTIONS:
Diagnostic Test: Chest X-ray Tomosynthesis — An imaging device that uses X-rays projected from multiple angles to reconstruct a three-dimensional images of the chest
  Other Names: CXRT

SUMMARY:
The goal of this observational clinical trial is to learn if chest tomosynthesis is a potential alternative to computed tomography for the detection of lung cancer. It will also develop artificial intelligence tools to aid in the diagnosis of lung cancer on chest tomosynthesis images. The main questions it aims to answer are:

* What is the accuracy of chest X-ray tomosynthesis in diagnosing lung cancer in a population of individuals undergoing lung cancer screening or evaluation of a suspicious lung nodule?
* Can artificial intelligence help us detect lung cancer on chest tomosynthesis images?

Researchers will compare chest tomosynthesis images to computed tomography scans for each participant to see how they compare in diagnosing lung cancer.

Participants will a chest tomosynthesis scan in addition to their routine clinical computed tomography scan.

DETAILED DESCRIPTION:
Lung cancer remains the most common cause of cancer death in the United States for which low-dose CT has proven benefit for early detection and survival from lung cancer. However, adoption remains low. Furthermore, >95% of nodules detected on low-dose CT, especially those smaller than 6 mm, do not represent cancer. We have partnered to develop a novel chest x-ray tomosynthesis (CXRT) device with the hypothesis that this device might be an alternative to CT for detection of lung cancer. We seek to recruit a cohort of patients to undergo CXRT, composed of patients concurrently undergoing lung cancer screening CT and diagnostic CT for new lung cancer. We will determine the effectiveness of CXRT for detecting lung cancer in this population, evaluating its sensitivity and specificity for detecting cancer and lung nodules at multiple size thresholds in a multireader study. We will additionally develop artificial intelligence algorithms and evaluate their efficacy to further enhance cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* undergoing lung cancer screening
* undergoing evaluation of suspicious pulmonary nodule
* newly diagnosed lung cancer

Exclusion Criteria:

* prior history of lung cancer treatment

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lung cancer screening CT or undergoing diagnostic chest CT for incidentally detected pulmonary nodules or lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Chest X-ray tomosynthesis detection of lung cancer | through 12/31/2026
  Diagnostic accuracy of chest tomosynthesis in identifying biopsy-proven lung cancer

SECONDARY OUTCOMES:
Chest X-ray tomosynthesis detection of suspicious nodules | through 12/31/2026
  Diagnostic accuracy of chest tomosynthesis in identifying pulmonary nodules seen on chest CT at multiple minimum size thresholds: 6-mm, 8-mm, 10-mm

CONTACTS AND LOCATIONS:
Overall Officials: Albert Hsiao, MD PhD, Principal Investigator — UC San Diego, Department of Radiology
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AIxScan, Inc — https://www.aixscan.com